CLINICAL TRIAL: NCT04587570
Title: Injection of Platelet Rich Plasma and Autologous Fat Into the Thumb Carpometacarpal Joint for the Evaluation Their Potential Filling Effect in Patients With Osteoarthritis
Brief Title: Rhizarthrosis Study
Acronym: RHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHI01
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Rhizarthrosis
Keywords: Rhizarthrosis
MeSH Terms: interventions — CD36 Antigens

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: Infiltration of PRP (Experimental): The proband gets Platelet Rich Plasma injected in the thumb saddle joint.
  Interventions: Procedure: Infiltration with PRP
- Group 2: Infiltration of Fat (Experimental): The proband gets fat injected in the thumb saddle joint.
  Interventions: Procedure: Infiltration with Fat
- Group 3: Infiltration of PRP and Fat (Experimental): The proband gets a mixture of Platelet Rich Plasma (PRP) and Fat injected in the thumb saddle joint.
  Interventions: Procedure: Infiltration with PRP and Fat
- Group 4: Infiltration of NaCl (Placebo Comparator): The proband gets NaCl injected in the thumb saddle joint.
  Interventions: Procedure: Infiltration with NaCl

INTERVENTIONS:
Procedure: Infiltration with PRP — Infiltration with 1.5 ml PRP
  Arms: Group 1: Infiltration of PRP
Procedure: Infiltration with Fat — Infiltration with 1.5 ml Fat
  Arms: Group 2: Infiltration of Fat
Procedure: Infiltration with PRP and Fat — Infiltration with 0.75 ml PRP and 0.75 ml Fat
  Arms: Group 3: Infiltration of PRP and Fat
Procedure: Infiltration with NaCl — Infiltration with 1.5 ml NaCl
  Arms: Group 4: Infiltration of NaCl

SUMMARY:
Rhizarthrosis is the wear of the thumb saddle joint. It is a very common disease affecting up to 25% of postmenopausal women. There are currently various conservative and surgical methods available for treatment. If conservative treatment does not lead to freedom from pain, one of the surgical methods can be used, such as metacarpal extension osteotomy, trapeziectomy with or without ligamentoplasty, trapeziometacarpal arthrodesis, prosthesis implantation and various forms of interposition arthroplasty . Despite the high satisfaction rate of up to 95% after surgical treatment, the anatomy of the carpus is irreversibly destroyed . Apart from that, these operations are also associated with corresponding complications and post-operative immobilization of several weeks. Thus, a minimally invasive treatment method with a corresponding success rate would be of great advantage.

Hypothesis:

By infiltrating and filling the joint with Platelet-Rich Plasma (PRP), fat or a combination of both, the pain of rhizarthrosis can be reduced.

Aim of the study:

The aim of the announced doctoral thesis is to investigate the effect of PRP, lipofilling and its combination on arthroses of the thumb saddle joint after a single joint injection and to compare it with a control group.It is to be proven that PRP, fat and their combination lead to a different degree of pain relief compared to the control group due to the expansion of the joint space and the associated filling effect.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed Rhizarthrosis

Exclusion Criteria:

* pregnancy and breastfeeding
* no signed Informed Consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Change in perception of pain sensation in the thumb saddle joint | is measured 5 times, from screening visit to 3 months after intervention
  assessed by VAS (Visual Analogue scale). The range goes from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in force in the thumb saddle joint. | is measured 5 times, from screening visit to 3 months after intervention.
  Evaluated by dynamometer: tweezergrip with Pinch-Gauge-Dynamometer, Crossgrip with Jamar-Dynamometer
Change in mobility of the thumb | is measured 5 times, from screening visit to 3 months after intervention.
  assessed by Kapandji-score, measured degrees of motion Dig I MCP, Dig I IP. A score of 0 indicates no opposition, a score of 10 indicates maximal opposition.
Change in quality of life score, assessed by Questionnaire SF36 | is measured 5 times, from screening visit to 3 months after intervention.
  The SF36 consists of 8 domains, the range of every scale goes from 0-100. A higher score indicates no restriction in health. 0 =greatest possible restriction of health; 100 = absence of health restrictions
Change in Disabilities of Arm, Shoulder and Hand (DASH) Score | is measured 5 times, from screening visit to 3 months after intervention.
  Upper-extremity disability and symptoms are assessed by the DASH-Score. The range goes from 0 (no disability) to 100.
Change in Michigan Hand Outcomes Questionnaire (MHQ) | is measured 5 times, from screening visit to 3 months after intervention.
  The MHQ has six domains. Overall hand function, activities of daily living (ADLs), work performance, aesthetics, and patient satisfaction) are scored from 0 - 100 in which 100 is the best possible ability.
  The pain domain is scored from 0 - 100, where 0 indicates no pain.
Change in movement in the thumb saddle joint. | is measured 5 times, from screening visit to 3 months after intervention.
  lateralgrip of dump and index finger

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Peter Kamolz, Univ. Prof. Dr., Principal Investigator — Medical University Graz, Department of Plastic, Aesthetic and Reconstructive Surgery; Raimund Winter, Dr., Principal Investigator — Medical University Graz, Department of Plastic, Aesthetic and Reconstructive Surgery
Locations (1):
- Medical University Graz, Department of Plastic, Aesthetic and Reconstructive Surgery Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No